CLINICAL TRIAL: NCT07127354
Title: The Impact of GLP-1 Agonist and GIP Agonist on Bowel Preparation Quality: A Randomized Controlled Trial
Brief Title: The Impact of GLP Medication on Colonoscopy Bowel Preparation Quality
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Shah,Tilak, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25-509
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: GLP - 1; Bowel Preparation for Colonoscopy
Keywords: GLP-1; Bowel preparation for colonoscopy

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Continue GLP/GIP medication (Active Comparator): Patient maintains dose, frequency, duration of medication prior to colonoscopy.
  Interventions: Drug: Continue GLP/GIP
- Hold medication (No Intervention): Withholds prior dose of GLP-1 or GIP therapy per ASA guidance recommendations

INTERVENTIONS:
Drug: Continue GLP/GIP — Continue GLP-1 or GIP-based therapy as prescribed prior to the procedure.
  Arms: Continue GLP/GIP medication

SUMMARY:
The goal of this clinical trial is to learn how GLP-1 and GIP agonists effect bowel preparation in patients scheduled for colonoscopies. The main questions it aims to answer are:

* Does GLP-1 and GIP agonist increase the rate of inadequate bowel preparation?
* Does the quality of bowel preparation differ in patients who hold vs. those who continue a single dose of their GLP-1 or GIP agonist medication?
* Are there any differences in the rates of complications gastric aspiration in patients who hold vs. continue a single dose of their GLP-1 or GIP agonist medication?

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (Age 18 years or older)
* Patient scheduled for outpatient screening, surveillance, or diagnostic colonoscopy
* Using a GLP-1 or GIP agonist at a stable dose for at least one month

Exclusion Criteria:

* Unable to provide informed consent, e.g., dementia
* Patient refuses the USMSTF recommended bowel cleansing regimen for patients with diabetes or obesity (split-dose 4 liters polyethylene glycol + 15 mg bisacodyl the afternoon before; low residue diet 3 days before colonoscopy; clear liquid diet the day before colonoscopy)
* Risk factors for inadequate bowel preparation besides diabetes and obesity with a likelihood ratio of 1.6 or greater:

  1. Cirrhosis
  2. Parkinson's disease
  3. Dementia
  4. Tricyclic antidepressant use
  5. Opioid use
  6. Gastroparesis* or suspected gastric outlet obstruction on pre-procedure imaging (*defined based on a documented 4-hour solid phase gastric emptying study or prior history of retained gastric contents during upper endoscopy)
  7. Previous colorectal surgery
  8. Prior history of inadequate bowel preparation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Rate of inadequate bowel preparation | During Surgery

SECONDARY OUTCOMES:
Median Boston bowel prep score | During Surgery
Median Ottawa bowel preparation score | During Surgery
Adenoma detection rate | During Surgery
Colonoscope Insertion time | During Surgery
  Time it takes to reach the cecum
Withdrawal time | During Surgery
Total procedure time | During Surgery
Rate of unplanned endotracheal intubation | During Surgery
hospitalization/emergency department evaluation/readmission for hypoxia or pnemonia within 96 hours after the procedure | From the day of the procedure to 96 hours after the procedure
Other serious adverse events | Day of the procedure up to 96 hours after the procedure.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cleveland Clinic, Cleveland, Florida
  - Cleveland Clinic Weston, Weston, Florida